CLINICAL TRIAL: NCT01391481
Title: The Randomized Controlled Trial (RCT) on the Vaporized Perfluorocarbon (PFC) Inhalation Treatment of Acute Respiratory Distress Syndrome With the Invasive Mechanical Ventilation（IMV）
Brief Title: Perfluorocarbon (PFC) Inhalation Treatment of Acute Lung Injury/Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The Second Artillery General Hospital (Other); The 306 Hospital of People's Liberation Army (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); General Hospital of Chinese Armed Police Forces (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Air Force General Hospital of the PLA (Other Government); 309th Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Principal Investigator, Chen Liang_An, M.D., Ph.D, Chinese PLA General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PLAGH-PFC
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Acute Lung Injury
Keywords: Perfluorocarbon; Acute Respiratory Distress Syndrome; Acute lung injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Fluorocarbons; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perfluorocarbon (Experimental)
  Interventions: Drug: Perfluorocarbon
- Sterile Water for Injection (Placebo Comparator)
  Interventions: Drug: Sterile Water for Injection

INTERVENTIONS:
Drug: Perfluorocarbon — Vaporized PFC Inhalation 100ml/8h for 5 days
  Arms: Perfluorocarbon
Drug: Sterile Water for Injection — Inhalation of Sterile Water for Injection, 100ml/8h for 5 days
  Arms: Sterile Water for Injection

SUMMARY:
PFCs (perfluorocarbons, PFC), an ideal liquid respiratory media, has special chemical and biological properties, including high solubility of gas, swiftness of carrying and release, low surface tension, high proportion, almost non-absorbing and non-metabolic characteristics in the body. On the basis of the strong animal data suggesting the efficacy of PFC vapor inhalation in models of lung injury, we performed a randomized clinical trial comparing PFC vapor inhalation with conventional mechanical ventilation（CMV）in patients with Acute Lung Injury/Acute Respiratory Distress Syndrome（ALI/ARDS）. The investigators will apply the Invasive Mechanical Ventilation (IMV) to the vaporized perfluorocarbon inhalation, objectively evaluate its curative effect on the acute respiratory distress syndrome, and meanwhile assess the safety of PFC.

DETAILED DESCRIPTION:
Based on the invasive mechanical ventilation (IMV) treatment of ALI/ARDS, the therapeutic action of vaporized PFC inhalation will be evaluated on the treatment of ALI/ARDS patients, and the safety of vaporized PFC inhalation on the treatment of ALI/ARDS. The Test group will make a timing and fix quantify inhalation of PFC, while the control group will be treated with the inhalation of water for injection. The general condition of patients will be assessed by monitoring their vital signs, hematology testing and APACHE II score, etc. Main outcome measures include the oxygenation index, respiratory mechanics; secondary outcomes include ventilator-free days, 28-day mortality and so on.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* Some clear risk aetiological agents of acute respiratory distress syndrome
* Acute onset, with corresponding clinical manifestations
* PaO2/FiO2 ≤ 300mmHg
* Chest radiograph or chest computerized tomography prompting bilateral pulmonary infiltrate shadow
* pulmonary capillary wedge pressure (PCWP) ≤ 18 mmHg or clinical cardiogenic pulmonary edema can be excluded
* respiratory rate (RR) ≥ 30bpm and (or) respiratory distress
* requiring tracheal intubation or tracheostomy for invasive mechanical ventilation
* or have received invasive mechanical ventilation time ≤ 3 days

Exclusion Criteria:

* Age: < 18 years old or > 75 years old
* During the early stage of the treatment, the use of mechanical ventilation for more than 3 days other than ALI/ARDS for reasons
* Lung parenchyma and airway surgery carried out within 30 days of the screening period
* Severe arrhythmia and myocardial ischemia after cardiopulmonary resuscitation
* Systolic blood pressure < 90 mm Hg, and can not maintain its stability with intravenous infusion and vasopressor drugs
* Intubation due to interstitial lung disease (E.g., sarcoidosis, idiopathic pulmonary fibrosis)
* Any active pneumothorax or mediastinal emphysema
* Risk factors leading to the death within 3 months in addition to ALI/ARDS during the screening period (E.g., end-stage cancer)
* Of perfluorocarbons' allergies
* Pregnant, breastfeeding women
* Attending other clinical trial within 30 days of the screening period
* Severe organ dysfunction (Marshall score ≥ 3 or Sequential Organ Failure Assessment（SOFA） score≥ 3, including serious liver and kidney dysfunction, upper gastrointestinal hemorrhage, etc.)
* Acute Physiology and Chronic Health Evaluation（APACHE） II score ≥ 30, high risk of death
* The researchers consider other situations not suitable for the case to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
oxygenation index, respiratory mechanics | three years
  oxygenation index and respiratory mechanics will be abtained before and 1, 2, 4h after every inhalation,

SECONDARY OUTCOMES:
Survival | three years
  ventilator-free days, 28-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Liangan Chen, M.D. PHD., Study Chair — Chinese PLA General Hospital
Locations (2):
- China (2):
  - 306 Hospital of PLA, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality